CLINICAL TRIAL: NCT03594994
Title: Metabolic Effects of Sleep Extension in People With Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 201805183; R01DK115502 (NIH)
Record Dates: First submitted 2018-06-28; First posted 2018-07-23 (Actual); Results first posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Insulin Resistance; Obesity
MeSH Terms: conditions — Insulin Resistance; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Maintain their usual sleep patterns
- Sleep Extension (Experimental): Extend sleep duration to >7h/night; 15 participants
  Interventions: Behavioral: Sleep extension

INTERVENTIONS:
Behavioral: Sleep extension — Extend time-in-bed by one hour
  Arms: Sleep Extension

SUMMARY:
This study is designed to determine the impact of extending sleep duration on glucose metabolism in people with obesity. Half of the participants will be instructed to increase their time-in-bed in order to achieve >7h sleep/night (sleep extension; n=15) while the other half will be be instructed to maintain their current sleep habits (n=15).

DETAILED DESCRIPTION:
Restricting sleep is known to be detrimental to glucose metabolism in healthy adults. Obesity is a condition associated with both lower sleep duration and poor glucose tolerance. Therefore, increasing sleep duration is a potentially novel therapeutic strategy for improving glucose metabolism in this population. The investigators will assess this by determining insulin sensitivity during a hyperinsulinemic-euglycemic clamp before and after a sleep intervention in both the control and sleep extension groups.

ELIGIBILITY:
Inclusion Criteria:

* Sleep <7h/night
* Body mass index 25-50 kg/m2
* Altered glucose metabolism (any of the following) Fasting glucose 100-125 mg/dL or, 2-h plasma glucose 140-199 mg/dL during an oral glucose tolerance test (OGTT) or, HbA1c 5.7-6.4% or, homeostatic model assessment of insulin resistance (HOMA-IR) ≥2.0

Exclusion Criteria:

* Sleep disorders

  1. moderate to severe sleep apnea (apnea-hypopnea index ≥15 events/hour)
  2. had ≥15 periodic limb movements per hour sleep [PLMS]
  3. narcolepsy or insomnia
* Perform shift work
* Excessive caffeine or alcohol consumption
* Significant organ dysfunction/disease (e.g. diabetes mellitus, kidney disease)
* Liver disease other than metabolic dysfunction associated steatotic liver disease (MASLD)
* Prior bariatric surgery
* Pregnancy or breastfeeding
* Taking medications that can affect study outcomes (alter sleep duration or glucose metabolism)
* Tobacco or illicit drug use
* Perform intense exercise >70 min/wk or moderate exercise >150 min/week
* Excessive alcohol consumption (>21 units of alcohol per week for men and >14 units of alcohol per week for women)

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 158 people were assessed for eligibility
Groups:
- Control: Maintain their usual sleep patterns; 16 participants
Period: Overall Study
Arm/Group | Control | Sleep Extension
Started | 16 | 15
Completed | 15 | 14
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Sleep Extension: Extend sleep duration to >7h/night
- Total: Total of all reporting groups
Arm/Group | Control | Sleep Extension | Total
Number analyzed (Participants) | 15 | 14 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (11) | 39 (13) | 41.8 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 22
  Male | 3 | 4 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White (Caucasian) | 8 | 7 | 15
  Black | 6 | 7 | 13
  Asian | 1 | 0 | 1
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 34.8 (5.6) | 35.5 (6.9) | 35.2 (6.2)
Fasting glucose [Mean (Standard Deviation); unit: mg/dL] | 94.9 (5.0) | 95.5 (4.1) | 95.2 (4.5)
120 min glucose [Mean (Standard Deviation); unit: mg/dL] — Measured during an oral glucose tolerance test, 120 minutes after ingesting a 75-g beverage
  mg/dL | 133 (29) | 127 (22) | 130.1 (25.4)
Homeostatic model assessment of insulin resistance [Mean (Standard Deviation); unit: 22.5/(µU/mL * mmol/L)] — The homeostasis model assessment of insulin resistance (HOMA-IR) was calculated by dividing the product of the plasma concentrations of insulin (in µU/mL) and glucose (in mmol/L) by 22.5. Higher values indicate greater insulin resistance.
  22.5/(µU/mL * mmol/L) | 4.3 (2.3) | 4.6 (2.3) | 4.4 (2.3)
Hemoglobin A1c [Mean (Standard Deviation); unit: %] | 5.4 (0.3) | 5.4 (0.5) | 5.4 (0.4)
Total sleep time [Mean (Standard Deviation); unit: hours] — Measured using wrist actigraphy
  hours | 6.1 (0.5) | 5.8 (0.5) | 6.0 (0.5)

OUTCOME MEASURES:

1. Primary Outcome: Insulin Sensitivity
Description: Whole-body insulin sensitivity calculated as the insulin stimulated rate of glucose disposal per kilogram of fat-free body mass (µmol/kgFFM/min) during a hyperinsulinemic-euglycemic clamp.
Time Frame: Change from baseline testing after 4-6 weeks of intervention
Measure: Mean (95% Confidence Interval); unit: µmol/kgFFM/min
Arm/Group | Control | Sleep Extension
Number analyzed (Participants) | 15 | 14
µmol/kgFFM/min | -3.8 [-8.6 to 0.9] | 0.9 [-5.0 to 6.8]

2. Secondary Outcome: Hepatic Insulin Sensitivity Index
Description: Calculated as the inverse of the product of plasma insulin concentration and endogenous glucose rate of appearance (Ra)/kgFFM during the basal period of the clamp procedure. Higher values indicate greater insulin sensitivity.
Time Frame: Change from baseline testing after 4-6 weeks of intervention
Measure: Mean (95% Confidence Interval); unit: 1000/[(µIU/mL) * (µmol/kg FFM/min)]
Arm/Group | Control | Sleep Extension
Number analyzed (Participants) | 15 | 14
1000/[(µIU/mL) * (µmol/kg FFM/min)] | 0.4 [-0.3 to 1.0] | -0.3 [-1.1 to 0.5]

3. Secondary Outcome: Adipose Tissue Insulin Sensitivity Index
Description: Calculated as the reciprocal of the product of palmitate Ra/kgFFM and plasma insulin concentration during basal conditions. Higher values indicate greater insulin sensitivity.
Time Frame: Change from baseline testing after 4-6 weeks of intervention
Measure: Mean (95% Confidence Interval); unit: 1000/[(µIU/mL) * (µmol/kg FFM/min)]
Arm/Group | Control | Sleep Extension
Number analyzed (Participants) | 13 | 14
1000/[(µIU/mL) * (µmol/kg FFM/min)] | 2.4 [-2.4 to 7.2] | -2.0 [-5.6 to 1.7]

4. Secondary Outcome: Homeostatic Model Assessment of Insulin Resistance
Description: The homeostasis model assessment of insulin resistance (HOMA-IR) was calculated by dividing the product of the plasma concentrations of insulin (in µU/mL) and glucose (in mmol/L) by 22.5. Higher values indicate greater insulin resistance.
Time Frame: Change from baseline testing after 4-6 weeks of intervention
Measure: Mean (95% Confidence Interval); unit: 22.5/(µU/mL * mmol/L)
Arm/Group | Control | Sleep Extension
Number analyzed (Participants) | 15 | 14
22.5/(µU/mL * mmol/L) | 0.2 [-0.6 to 0.9] | 0.3 [-0.7 to 1.2]

5. Secondary Outcome: 24 Hour Glucose Area Under the Concentration Curve
Description: Plasma metabolite concentrations will be evaluated over a 24 hour period
Time Frame: Change from baseline testing after 4-6 weeks of intervention
Measure: Mean (95% Confidence Interval); unit: mg/dL x 24 h
Arm/Group | Control | Sleep Extension
Number analyzed (Participants) | 13 | 12
mg/dL x 24 h | 45 [0 to 90] | 41 [-23 to 105]

6. Secondary Outcome: 24 Hour Insulin Area Under the Concentration Curve
Description: Plasma insulin concentrations evaluated over a 24 hour period
Time Frame: Change from baseline testing after 4-6 weeks of intervention
Measure: Mean (95% Confidence Interval); unit: mU/L x 24 h
Arm/Group | Control | Sleep Extension
Number analyzed (Participants) | 13 | 12
mU/L x 24 h | 1 [-196 to 197] | -44 [-197 to 109]

7. Secondary Outcome: 24 Hour Non-esterified Fatty Acids Area Under the Concentration Curve
Description: Plasma metabolite concentrations will be evaluated over a 24 hour period
Time Frame: Change from baseline testing after 4-6 weeks of intervention
Measure: Mean (95% Confidence Interval); unit: mg/dL x 24 h
Arm/Group | Control | Sleep Extension
Number analyzed (Participants) | 13 | 12
mg/dL x 24 h | 1.0 [0.1 to 2.0] | -0.3 [-1.3 to 0.7]

8. Secondary Outcome: Body Mass
Description: Measured using a body weight scale
Time Frame: Change from baseline testing after 4-6 weeks of intervention
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | Control | Sleep Extension
Number analyzed (Participants) | 15 | 14
kg | -1.1 [-2.5 to 0.3] | -0.3 [-1.1 to 0.5]

9. Secondary Outcome: Fat-free Mass
Description: Body composition assessed using dual-energy x-ray absorptiometry (DXA)
Time Frame: Change from baseline testing after 4-6 weeks of intervention
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | Control | Sleep Extension
Number analyzed (Participants) | 15 | 14
kg | -0.2 [-1.1 to 0.7] | -0.5 [-1.6 to 0.7]

10. Secondary Outcome: Body Fat
Description: Body composition assessed using dual-energy x-ray absorptiometry (DXA)
Time Frame: Change from baseline testing after 4-6 weeks of intervention
Measure: Mean (95% Confidence Interval); unit: % of total body mass
Arm/Group | Control | Sleep Extension
Number analyzed (Participants) | 15 | 14
% of total body mass | 0.5 [-0.1 to 1.2] | 0.4 [-0.2 to 1.0]

11. Secondary Outcome: Liver Fat
Description: Proton-density fat fraction of the whole liver assessed by using magnetic resonance imaging (MRI)
Time Frame: Change from baseline testing after 4-6 weeks of intervention
Measure: Mean (95% Confidence Interval); unit: % of whole liver
Arm/Group | Control | Sleep Extension
Number analyzed (Participants) | 15 | 14
% of whole liver | -0.63 [-2.01 to 0.76] | 0.6 [-0.04 to 1.26]

12. Secondary Outcome: Fasting Glucose
Description: Plasma glucose measured after an overnight fast
Time Frame: Change from baseline testing after 4-6 weeks of intervention
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Control | Sleep Extension
Number analyzed (Participants) | 15 | 14
mg/dL | 3.6 [0.6 to 6.7] | 0.8 [-2.2 to 3.8]

13. Secondary Outcome: Daily Time in Bed
Description: Assessed by using actigraphy over 7 days
Time Frame: Change from baseline testing after 4-6 weeks of intervention
Measure: Mean (95% Confidence Interval); unit: hours
Arm/Group | Control | Sleep Extension
Number analyzed (Participants) | 15 | 14
hours | 0.3 [-0.2 to 0.7] | 1.3 [1.0 to 1.7]

14. Secondary Outcome: Daily Total Sleep Time
Description: Assessed by using actigraphy over 7 days
Time Frame: Change from baseline testing after 4-6 weeks of intervention
Measure: Mean (95% Confidence Interval); unit: hours
Arm/Group | Control | Sleep Extension
Number analyzed (Participants) | 15 | 14
hours | 0.0 [-0.2 to 0.2] | 1.1 [0.8 to 1.4]

15. Secondary Outcome: Stage N1 Sleep Time
Description: Assessed by using inpatient polysomnography
Time Frame: Change from baseline testing after 4-6 weeks of intervention
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Control | Sleep Extension
Number analyzed (Participants) | 13 | 10
minutes | -1.3 [-5.9 to 3.2] | 6.9 [-1.6 to 15.3]

16. Secondary Outcome: Stage N2 Sleep Time
Description: Assessed by using inpatient polysomnography
Time Frame: Change from baseline testing after 4-6 weeks of intervention
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Control | Sleep Extension
Number analyzed (Participants) | 13 | 10
minutes | -11.7 [-52.3 to 28.9] | 23.9 [11.8 to 59.6]

17. Secondary Outcome: Stage N3 Sleep Time
Description: Assessed by using inpatient polysomnography
Time Frame: Change from baseline testing after 4-6 weeks of intervention
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Control | Sleep Extension
Number analyzed (Participants) | 13 | 10
minutes | 4.4 [-12.1 to 21.0] | 14.9 [-2.6 to 32.4]

18. Secondary Outcome: Rapid Eye Movement (REM) Sleep Time
Description: Assessed by using inpatient polysomnography
Time Frame: Change from baseline testing after 4-6 weeks of intervention
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Control | Sleep Extension
Number analyzed (Participants) | 13 | 10
minutes | -1.6 [-16.0 to 12.8] | 7.6 [-21.9 to 37.0]

ADVERSE EVENTS:
Time Frame: Before, during and after the 4-6 week intervention
Arm/Group | Control | Sleep Extension
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 1/16 | 0/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=16) | Sleep Extension (N=15)
Unrelated medical issue (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Broken foot during the a motorcycle accident during the habitual sleep intervention period

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-10-08): https://cdn.clinicaltrials.gov/large-docs/94/NCT03594994/Prot_SAP_000.pdf